CLINICAL TRIAL: NCT03159637
Title: Impact Of Posture and Prolonged Pneumoperitoneum on Intra-Operative and Postoperative Outcomes During Gynecological Laparoscopic Surgery: An Observational Clinical Study
Brief Title: Pneumoperitoneum and Gynecological Laparoscopic Surgery: An Observational Clinical Study
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Profossor, Assiut University
Other Study IDs: IRB000087698
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Laparoscopy
Keywords: Pneumoperitoneum; Trendelenburg position; intra-abdominal pressure
MeSH Terms: conditions — Pneumoperitoneum | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic Surgery — Insufflation of a gas (carbon dioxide) into the peritoneal cavity producing a pneumoperitoneum will be done. The positioning of the patients in Trendelenburg position will be done. intraoperative and postoperative outcomes will be assesed

SUMMARY:
Laparoscopic surgery is now widely established.Laparoscopic surgery involves insufflation of a gas (usually carbon dioxide) into the peritoneal cavity producing a pneumoperitoneum. The raised intra-abdominal pressure of the pneumoperitoneum, alteration in the patient's position and effects of carbon dioxide absorption cause changes in physiology, especially within the cardiovascular and respiratory systems.

DETAILED DESCRIPTION:
The study will be carried out after approval of the ethical committee of Faculty of Medicine, Assiut University. A full preoperative anesthetic assessment will be carried out. Particular attention to the cardiovascular and respiratory systems is essential because of potential effects of the pneumoperitoneum and patient position.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-50
2. ASA 1
3. Elective gynecological laparoscopic surgery

Exclusion Criteria:

1. Severe ischemic or valvular heart disease
2. Increased intracranial pressure (e.g. Hydrocephalus, Cerebral tumor, Head injury)
3. Hepatic or renal impairment
4. Emergency surgery
5. Open surgery
6. Previous abdominal surgery

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female patients only
Study Population: female patients only
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure | within the duration of the operation
  mean arterial blood pressure will be monitored at different times
Pulmonary function tests | within the first 24 hours
  forced expiratory volume at one second

SECONDARY OUTCOMES:
PaO2 | within the first 24 hours
  PaO2 will be monitored at different times
Arterial to end-tidal PaCO2- difference | within the first 24 hours
  Arterial to end-tidal PaCO2- difference will be monitored at different times
Intra-abdominal pressure | within the first 24 hours
  Intra-abdominal pressure by direct measurement and indirect by Foley´s catheter will be monitored at different times (Cm water)
Postoperative nausea and vomiting | within the first 24 hours
  Postoperative nausea and vomiting will be monitored at different times by special scale
Analgesic requirement | within the first 24 hours
  Analgesic requirement will be monitored at different times by special scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Sayed K Abd-Elshafy, M.D, Principal Investigator — Associate Profossor
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided